CLINICAL TRIAL: NCT06443502
Title: An Open-label Single-Arm Phase 3 Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Vedolizumab Intravenous in the Treatment of Pediatric Subjects With Active Chronic Pouchitis
Brief Title: A Study to Learn About the Safety of Vedolizumab and How Well it Works in Children and Teenagers With Active Chronic Pouchitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vedolizumab-3041; 2023-504773-20-00 (EU CTIS Number: EU CT Number)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pouchitis
Keywords: Drug Therapy
MeSH Terms: conditions — Pouchitis | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vedolizumab (Experimental): Participants will receive vedolizumab intravenous infusion based on body weight (>=30 kg: high dose, >15 to <30 kg: medium dose, 10-15 kg: low dose) on Day 1, Weeks 2 and 6 during induction period and every 8 weeks (Q8W) at Weeks 14, 22 and 30 during maintenance period. Ciprofloxacin, metronidazole, vancomycin, amoxicillin-clavulanate, or rifaximin, will be administered as concomitant antibiotics, orally from Day 1 to Week 2 during induction period (unless intolerant or contraindicated) in Part 1. Participants who respond at Week 34 will proceed to Part 2 and will continue to receive vedolizumab intravenous infusions every 8 weeks from Week 38 to Week 78 throughout continued maintenance Part 2. The dose of vedolizumab used during Part 2 will be the same as the last dose administered during Week 30 of Part 1.
  Interventions: Drug: Vedolizumab; Drug: Concomitant Antibiotic Therapy

INTERVENTIONS:
Drug: Vedolizumab — Vedolizumab intravenous infusion.
  Other Names: Entyvio; MLN0002; Kynteles
Drug: Concomitant Antibiotic Therapy — Ciprofloxacin, metronidazole, vancomycin, amoxicillin clavulanate or rifaximin.

SUMMARY:
When some people have their large bowel removed, a surgeon can make a "pouch" from part of the small bowel to connect it to the back passage (anus). Pouchitis is when the pouch becomes inflamed (swollen) or infected. The main aim of this study is to find out if vedolizumab improves pouchitis symptoms and pouch inflammation. Other aims include to find out if vedolizumab is well tolerated and if it causes any medical problems (adverse events or side effects) and to look for any changes in the well-being of participants during their treatment with vedolizumab.

This study consists of two parts: Part 1 includes the induction and maintenance periods, and Part 2 includes the continued maintenance period. Participants will receive up to 12 infusions of vedolizumab. In Part 1 of the study, first 3 infusions are in first 6 weeks (Day 1, Week 2 and Week 6). Participants who are getting benefit may continue with the treatment for up to 7.5 months (30 weeks) in the maintenance period for Part 1. After completing treatment with vedolizumab in Part 1, participants will visit their clinic for a health check at Week 34.

Participants who show clinical response at Week 34 will continue to Part 2, receiving vedolizumab every 8 weeks for an additional 40 weeks, starting at Week 38 and ending with the last dose being at Week 78. Final efficacy assessments, including a pouchoscopy will be performed at Week 82.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab. This study will look at the efficacy, safety, tolerability, pharmacokinetics (PK), and immunogenicity of vedolizumab in pediatric participants with active chronic pouchitis.

The study will enroll approximately 30 participants. All the participants will be enrolled in a single treatment group to receive treatment with vedolizumab based on participant's weight mentioned as follows:

* Participants with body weight greater than or equal to (>=) 30 kilogram (kg) will receive vedolizumab, high dose
* Participants with body weight greater than (>) 15 to less than (<) 30 kg will receive vedolizumab, medium dose
* Participants with body weight 10 to 15 kg will receive vedolizumab, low dose

All participants will receive vedolizumab intravenous infusion at Day 1, and at Weeks 2, 6, 14, 22, and 30. Participants will also receive concomitant antibiotic treatment (ciprofloxacin, metronidazole, or other antibiotics) from Day 1 through Week 2. Participants with clinical response at the end of Part 1 maintenance at Week 34 will continue to Part 2 of the study and will receive vedolizumab intravenous infusion every 8 weeks from Week 38 through Week 78.

This multi-center trial will be conducted globally. The maximum overall duration of the study is up to approximately 2 years. Participants will be followed up for 18 weeks after the last dose of the study drug for safety.

ELIGIBILITY:
Inclusion Criteria:

1. The participant weighs >=10 kg at the time of screening and first dose.
2. Has active chronic pouchitis, defined by a mPDAI score >=5 assessed using the 3-day average of participant-reported clinical symptoms prior to the screening endoscopy (that is [ie] video pouchoscopy with biopsy) or bowel preparation for the endoscopy and a minimum mPDAI endoscopic subscore of 2 (outside the staple or suture line) and either:

   * >=1 previous episodes of pouchitis within 1 year before the screening visit, with symptoms lasting for at least a total of 4 weeks, treated with >=2 weeks of antibiotic or other prescription therapy (ie, other antibiotics, probiotics, immunomodulators, or anti-tumor necrosis factor [TNFs] within 1 year before screening). Or
   * Have had an inadequate response with, or lost response to, or be intolerant to antibiotic therapy (ie, requiring maintenance antibiotic therapy taken for >=4 weeks immediately before the baseline endoscopy visit or not able to receive or continue antibiotic treatment due to intolerance or other contraindication).
3. The participant is aged 2 to 17 years, inclusive, at the time of screening and first dose.
4. The participant has a history of proctocolectomy and ileal pouch-anal anastomosis (IPAA) as treatment for ulcerative colitis (UC), Crohn's disease (CD), familial adenomatous polyposis (FAP), or other underlying conditions, such as Hirschsprung's disease, for which construction of a pouch was medically indicated, completed at least 1 year before the screening visit.

Exclusion Criteria:

The exclusion criteria are divided into 3 categories: active chronic pouchitis exclusion criteria, infectious disease exclusion criteria, and general exclusion criteria.

Active Pouchitis Exclusion Criteria:

1. Has symptoms believed to be predominantly due to irritable pouch syndrome.
2. Has isolated cuffitis.
3. Is found to have dysplasia at the screening endoscopy.
4. Has mechanical complications of the pouch (for example [e.g.] pouch stricture or pouch fistula).
5. Currently requires or has a planned surgical intervention during the study.
6. Has a diverting stoma.

   Infectious Disease Exclusion Criteria:
7. Has evidence of an active infection (e.g. sepsis, cytomegalovirus [CMV], or listeriosis) during screening.
8. Had a clinically significant infection (e.g. pneumonia, pyelonephritis, coronavirus disease 2019 [COVID-19]) within 35 days before first dose of study drug.
9. Has active or latent tuberculosis (TB), as evidenced by a diagnostic TB test performed within 3 months of screening or during the screening period that is positive, as defined by:

   * A positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, or
   * A TB skin test reaction >=5 millimeter (mm). NOTE: If participant have received Bacillus Calmette-Guérin vaccine, then a QuantiFERON TB Gold test should be performed instead of the TB skin test.

   NOTE: Participants with documented previously treated TB with a negative QuantiFERON test can be included in the study.
10. Has evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Hepatitis B virus (HBV) immune participants (e.g. HBsAg negative and hepatitis B antibody positive) may, however, be included.

    NOTE: If a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if the absence of HBV DNA is confirmed by HBV DNA polymerase chain reaction reflex testing performed in the central laboratory.
11. Has chronic hepatitis C virus (HCV) (ie, positive HCV antibody [HCVAb] and HCV Ribonucleic Acid [RNA]).

    NOTE: Participants who are HCVAb-positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks before baseline]).
12. Has any identified congenital or acquired immunodeficiency (e.g. common variable immunodeficiency, HIV infection, organ transplantation).
13. Has positive stool studies for ova and/or parasites or stool culture at screening visit.
14. Has positive Clostridium difficile stool test at screening visit.

    General Exclusion Criteria:
15. Is taking, has taken, or is required to take any excluded medications.
16. Has active cerebral/meningeal disease, signs/symptoms, or history of progressive multifocal leukoencephalopathy (PML) or any other major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
17. Has evidence of dysplasia or history of malignancy other than a successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix.
18. Has any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, GI, genitourinary, hematologic, coagulation, immunological, endocrine/metabolic, neurologic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise participant safety.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Modified Pouchitis Disease Activity Index (mPDAI) Remission at Week 14 | At Week 14
  Clinical (mPDAI) remission is defined as mPDAI score <5 and a reduction of mPDAI score by >=2 points from Baseline. The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees celsius [C]) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical (mPDAI) Remission at Week 34 | At Week 34
  Clinical (mPDAI) remission is defined as mPDAI score <5 and a reduction of mPDAI score by >=2 points from Baseline. The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees C) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.
Percentage of Participants Achieving Pouchitis Disease Activity Index (PDAI) Remission at Week 14 | At Week 14
  PDAI remission is PDAI score <7 and reduction of score by >=3 points from Baseline. PDAI score calculated as sum of 3 subscales based on clinical symptoms (0-6), endoscopic findings (EF) (0-6), and histologic changes (0-6): 1)Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare,1=Present daily); Fecal urgency or abdominal cramps (0=None, 2=Usual),Fever (temperature>37.8 degree C) (0=Absent,1=Present);2) EF Findings: Edema (0=not present, 1=present);Granularity (0=not present, 1=present); Friability (0=not present,1=present);Loss of vascular pattern (0=not present, 1=present); Mucous exudates (0=not present, 1=present);Ulcerations (0=not present,1=present);3) Acute Histologic Inflammation: Polymorphic nuclear leukocyte infiltration (0=None, 3=Severe+crypt abscess); Ulceration per low power field (mean) (0=0% to 3=>50%). Total PDAI score ranges 0-18. Higher score means worse disease.
Percentage of Participants Achieving PDAI Remission at Week 34 | At Week 34
  PDAI remission is PDAI score <7 and reduction of score by >=3 points from Baseline. PDAI score calculated as sum of 3 subscales based on clinical symptoms (0-6), EF (0-6), and histologic changes (0-6): 1)Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare,1=Present daily); Fecal urgency or abdominal cramps (0=None, 2=Usual),Fever (temperature>37.8 degree C) (0=Absent,1=Present);2) EF Findings: Edema (0=not present, 1=present);Granularity (0=not present, 1=present); Friability (0=not present,1=present);Loss of vascular pattern (0=not present, 1=present); Mucous exudates (0=not present, 1=present);Ulcerations (0=not present,1=present);3) Acute Histologic Inflammation: Polymorphic nuclear leukocyte infiltration (0=None, 3=Severe+crypt abscess); Ulceration per low power field (mean) (0=0% to 3=>50%). Total PDAI score ranges 0-18. Higher score means worse disease.
Percentage of Participants Achieving Clinical (mPDAI) Response at Week 14 | At Week 14
  Clinical (mPDAI) response is defined as a reduction in mPDAI score by >=2 points from baseline. The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees C) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.
Percentage of Participants Achieving Clinical (mPDAI) Response at Week 34 | At Week 34
  Clinical (mPDAI) response is defined as a reduction in mPDAI score by >=2 points from baseline. The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees C) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.
Change From Baseline in (mPDAI) Total Score at Week 14 | Baseline, Week 14
  The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees C) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.
Change From Baseline in (mPDAI) Total Score at Week 34 | Baseline, Week 34
  The mPDAI score is calculated as a sum of two subscales based on clinical symptoms (0 to 6) and endoscopic findings (0 to 6): 1) Clinical Symptoms: Stool Frequency (0=usual postoperative stool frequency to 2=three or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature >37.8 degrees C) (0=Absent and 1=Present); 2) Endoscopic Inflammation Findings: Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). The total mPDAI score can range from 0 to 12. A higher mPDAI score is indicative of worse disease.
Change From Baseline in PDAI Total Score at Week 14 | Baseline, Week 14
  The PDAI score calculated as sum of 3 subscales based on clinical symptoms (0-6), endoscopic findings (0-6), and histologic changes (0-6): 1)Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare,1=Present daily); Fecal urgency or abdominal cramps (0=None, 2=Usual),Fever (temperature>37.8 degree C) (0=Absent,1=Present); 2) Endoscopic Findings: Edema (0=not present, 1=present);Granularity (0=not present, 1=present); Friability (0=not present,1=present);Loss of vascular pattern (0=not present, 1=present); Mucous exudates (0=not present, 1=present);Ulcerations (0=not present,1=present);3) Acute Histologic Inflammation: Polymorphic nuclear leukocyte infiltration (0=None, 3=Severe + crypt abscess); Ulceration per low power field (mean) (0=0 percentage [%] to 3=>50%). Total PDAI score ranges from 0-18. Higher score means worse disease.
Change From Baseline in PDAI Total Score at Week 34 | Baseline, Week 34
  The PDAI score calculated as sum of 3 subscales based on clinical symptoms (0-6), endoscopic findings (0-6), and histologic changes (0-6): 1)Clinical Symptoms: Stool Frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare,1=Present daily); Fecal urgency or abdominal cramps (0=None, 2=Usual),Fever (temperature>37.8 degree C) (0=Absent,1=Present); 2) Endoscopic Findings: Edema (0=not present, 1=present);Granularity (0=not present, 1=present); Friability (0=not present,1=present);Loss of vascular pattern (0=not present, 1=present); Mucous exudates (0=not present, 1=present);Ulcerations (0=not present,1=present);3) Acute Histologic Inflammation: Polymorphic nuclear leukocyte infiltration (0=None, 3=Severe + crypt abscess); Ulceration per low power field (mean) (0=0 percentage [%] to 3=>50%). Total PDAI score ranges from 0-18. Higher score means worse disease.
Change From Baseline in PDAI Clinical Symptoms Subscore at Week 14 | Baseline, Week 14
  The PDAI Clinical Symptoms subscore is a sum of scores (0 to 6) from findings for stool frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature>37.8 degree C) (0=Absent to 1=Present). Higher scores are indicative of worse disease.
Change From Baseline in PDAI Clinical Symptoms Subscore at Week 34 | Baseline, Week 34
  The PDAI Clinical Symptoms subscore is a sum of scores (0 to 6) from findings for stool frequency (0=usual to postoperative stool frequency to 2=3 or more stools/day>postoperative usual); Rectal bleeding (0=None or rare to 1=Present daily); Fecal urgency or abdominal cramps (0=None to 2=Usual), Fever (temperature>37.8 degree C) (0=Absent to 1=Present). Higher scores are indicative of worse disease.
Change From Baseline in PDAI Endoscopic Subscore at Week 14 | Baseline, Week 14
  The PDAI Endoscopic Inflammation subscore is a sum of scores (0 to 6) from findings for Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). Higher scores are indicative of worse disease.
Change From Baseline in PDAI Endoscopic Subscore at Week 34 | Baseline, Week 34
  The PDAI Endoscopic Inflammation subscore is a sum of scores (0 to 6) from findings for Edema (0=not present to 1=present); Granularity (0=not present to 1=present); Friability (0=not present to 1=present); Loss of vascular pattern (0=not present to 1=present); Mucous exudates (0=not present to 1=present); Ulcerations (0=not present to 1=present). Higher scores are indicative of worse disease.
Change From Baseline in PDAI Acute Histologic Inflammation Subscore at Week 14 | Baseline, Week 14
  The PDAI Acute Histologic Inflammation subscore is a sum score (0 to 6) from findings for Polymorphic nuclear leukocyte infiltration (0=None to 3=Severe + crypt abscess); Ulceration per low power field (mean) (0=0% to 3=>50%). Higher scores are indicative of worse disease.
Change From Baseline in PDAI Acute Histologic Inflammation Subscore at Week 34 | Baseline, Week 34
  The PDAI Acute Histologic Inflammation subscore is a sum score (0 to 6) from findings for Polymorphic nuclear leukocyte infiltration (0=None to 3=Severe + crypt abscess); Ulceration per low power field (mean) (0=0% to 3=>50%). Higher scores are indicative of worse disease.
EuroQol- 5 Dimension for Youth (EQ-5D-Y) Index Scores and Visual Analogue Scale (VAS) at Week 14 | At Week 14
  The EQ-5D-Y (Proxy Version 1.0) is composed of two sections. The first section contains one question for each of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. Participants select from three response levels (no problems, some problems, a lot of problems) for each dimension. A health state profile score can be calculated from the responses on these five dimensions. The index score ranges from 0 (0 indicating a health state equivalent to death) to 1 (indicating full health). Higher scores demonstrate higher health utility. The second section includes a VAS (EuroQol [EQ] VAS). The scale is scored from 0 (the worst) to 100 (the best imaginable health). The reference to a high score indicates a better outcome of quality of life.
EQ-5D-Y Index Scores and VAS at Week 34 | At Week 34
  The EQ-5D-Y (Proxy Version 1.0) is composed of two sections. The first section contains one question for each of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. Participants select from three response levels (no problems, some problems, a lot of problems) for each dimension. A health state profile score can be calculated from the responses on these five dimensions. The index score ranges from 0 (0 indicating a health state equivalent to death) to 1 (indicating full health). Higher scores demonstrate higher health utility. The second section includes a VAS (EQ VAS). The scale is scored from 0 (the worst) to 100 (the best imaginable health). The reference to a high score indicates a better outcome of quality of life.
Change From Baseline in the EQ-5D-Y Index Scores and VAS at Week 14 | Baseline, Week 14
  The EQ-5D-Y (Proxy Version 1.0) is composed of two sections. The first section contains one question for each of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. Participants select from three response levels (no problems, some problems, a lot of problems) for each dimension. A health state profile score can be calculated from the responses on these five dimensions. The index score ranges from 0 (0 indicating a health state equivalent to death) to 1 (indicating full health). Higher scores demonstrate higher health utility. The second section includes a VAS (EQ VAS). The scale is scored from 0 (the worst) to 100 (the best imaginable health). The reference to a high score indicates a better outcome of quality of life.
Change From Baseline in the EQ-5D-Y Index Scores and VAS at Week 34 | Baseline, Week 34
  The EQ-5D-Y (Proxy Version 1.0) is composed of two sections. The first section contains one question for each of the five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad, or unhappy. Participants select from three response levels (no problems, some problems, a lot of problems) for each dimension. A health state profile score can be calculated from the responses on these five dimensions. The index score ranges from 0 (0 indicating a health state equivalent to death) to 1 (indicating full health). Higher scores demonstrate higher health utility. The second section includes a VAS (EQ VAS). The scale is scored from 0 (the worst) to 100 (the best imaginable health). The reference to a high score indicates a better outcome of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium
- Children's Hospital Zagreb, Zagreb, Croatia
- Fakultni nemocnice v Motole, Pediatricka klinika 2, Prague, Czechia
- Sotiria Thoracic Diseases Hospital, Dpt. of Gastroenterology, Building Z, Athens, Attica, Greece
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Italy (5):
  - Istituto G Gaslini Ospedale Pediatrico IRCCS, Genova
  - Azienda Ospedaliero Universitaria, Policlinico Gaetano Martino, Messina
  - AOU dell'Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Rome
  - IRCCS Materno Infantile Burlo Garofolo, Trieste
- Instytut Pomnik-/Centrum Zdrowia dziecka, Warsaw, Poland
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitari I Politecnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/01f2fb690a434210??page=1&idFilter=Vedolizumab-3041